CLINICAL TRIAL: NCT05758636
Title: The Effect of Emotional Freedom Technique on Anxiety Levels of Nurses Who Care for COVID19 Patients During the Pandemic Process
Brief Title: The Effect of Emotional Freedom Technique on Anxiety Levels of Nurses Caring for COVID19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, gulsah okut, Phd Candidate, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MrmrU
Record Dates: First submitted 2023-03-04; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: EFTs; Nursing Caries; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Freedom Technique Group (Experimental): Nurses (40) enrolled in the emotional freedom technique group will receive a total of 4 rounds of EFT, 50 minutes, 3 days a week.
  Interventions: Behavioral: Emotional Freedom Technique
- Control (No Intervention): Participants in the control group (n= 40) will not receive intervention throughout the study.

INTERVENTIONS:
Behavioral: Emotional Freedom Technique — Before starting the EFT session, the participants were asked to identify the problem that aroused their anxiety. After the common point of the problems was determined, the ORDS level of all participants was determined. Next, the EFT session explained traditional acupressure meridian points on the head, face, neck, chest, and hands. Next, they were asked to repeat the phrase, "Even though I have this feeling of stress and anxiety, I accept myself deeply and completely," while gently applying to the acupuncture points with their index and middle fingers. While using this expression, the participants hit each acupuncture area seven times. After the first round of hits accompanied by this phrase, participants were asked to abbreviate "this feeling of anxiety, stress" with another short phrase. The participants then repeated rounds of this process until they noticed that their anxiety had decreased
  Arms: Emotional Freedom Technique Group

SUMMARY:
It is very important to protect and improve the physical, mental and social health of nurses, especially in the event that nurses frequently encounter patients diagnosed or suspected of COVID-19 and are exposed to the virus for a long time due to the long duration of care, increasing cases and the death of their colleagues. Que et al., 2020). Current researches have made it necessary for nurses to have difficulties in effectively coping with the anxiety experienced in the COVID-19 pandemic, which has affected the whole world, and to apply new effective methods, as their training includes effective coping methods (Feinstein and Church, 2010). There are studies that are effective in reducing stress and anxiety, such as meditation, yoga, and breathing therapies, which are recommended to prevent the increase in stress and anxiety levels that may occur in nurses by evaluating the experienced situations (Labrague et al., 2020; Vieta et al., 2020). In addition to these applications, it is seen that Emotional Freedom Technique (EFT) has been increasingly used recently in controlling and reducing anxiety (Hartmann, 2016). EFT is a type of energy-based psychotherapy that combines the components of Western psychology and Eastern medicine, applied to eliminate negative thoughts and feelings and problems related to emotions (İnangil et al., 2020; Church, 2013). Although the EFT technique is used in many different areas today, its effect on the level of anxiety in nurses during the COVID-19 process is not yet known. As a result, to evaluate the effect of EFT, whose positive results have been proven by many studies, on the anxiety level of nurses caring for COVID-19 patients.

DETAILED DESCRIPTION:
It is very important to protect and improve the physical, mental and social health of nurses in the event that they are exposed to the virus for a long time due to the frequent encounters with patients diagnosed or suspected of COVID-19 and the long duration of care, increasing cases and the death of their colleagues (Que et al., 2020). Current researches have made it necessary for nurses to have difficulties in effectively coping with the anxiety experienced in the COVID-19 pandemic, which has affected the whole world, and to apply new effective methods, as their training includes effective coping methods (Feinstein and Church, 2010). It is very important to protect and improve the physical, mental and social health of nurses, especially in the event that nurses frequently encounter patients diagnosed or suspected of COVID-19 and are exposed to the virus for a long time due to the long duration of care, increasing cases and the death of their colleagues. Que et al., 2020). Current researches have made it necessary for nurses to have difficulties in effectively coping with the anxiety experienced in the COVID-19 pandemic, which has affected the whole world, and to apply new effective methods, as their training includes effective coping methods (Feinstein and Church, 2010). There are studies that are effective in reducing stress and anxiety, such as meditation, yoga, and breathing therapies, which are recommended to prevent the increase in stress and anxiety levels that may occur in nurses by evaluating the experienced situations (Labrague et al., 2020; Vieta et al., 2020). In addition to these applications, it is seen that Emotional Freedom Technique (EFT) has been increasingly used recently in controlling and reducing anxiety (Hartmann, 2016). EFT is a type of energy-based psychotherapy that combines the components of Western psychology and Eastern medicine, applied to eliminate negative thoughts and feelings and problems related to emotions (İnangil et al., 2020; Church, 2013). In the process of providing effective care to COVID-19 cases, nurses fulfill the requirements of their profession with their ability to anticipate some unforeseen problems created by the workplace environment and to solve these problems. Due to the challenging process that emerged with the pandemic, the treatment and care of their patients, as well as meeting many urgent needs, left nurses in a difficult situation (Labrague et al., 2020; Vieta et al., 2020). It is very important that nurses, who provide services effectively and in a competitive way during the pandemic, can protect their physical, mental and social health (Chirico et al., 2020). Although the EFT technique is used in many different areas today, its effect on the level of anxiety in nurses during the COVID-19 process is not yet known. As a result, to evaluate the effect of EFT, whose positive results have been proven by many studies, on the anxiety level of nurses caring for CO

ELIGIBILITY:
Inclusion Criteria:

* not having been diagnosed with a psychiatric diagnosis,
* not having received any therapy including coping with stress
* not being diagnosed with COVID-19
* not being in the treatment care process
* not having applied the emotional freedom technique before, and volunteering to participate

Exclusion Criteria:

* Not participating in any of the emotional freedom technique sessions
* Being diagnosed with COVID-19 during the application of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Spielberger state-trait anxiety scale | 4 months
  While the Trait Anxiety Inventory aims to determine how the individual feels independently of the situation and conditions, the State Anxiety Inventory aims to determine how the individual feels at a certain moment and under certain conditions. Both subscales are four-point Likert-type scales consisting of twenty items. In the State Anxiety Inventory, the individual is asked to evaluate how he or she feels at the moment, according to the situation he is in, and to choose one of the expressions "1-not at all, 2-somewhat, 3-a lot and 4-completely" according to the severity of the emotions or behaviors expressed in the items. The highest score of 4 is given for choosing the phrase "completely", and the lowest score is 1 for choosing the phrase "not at all".

SECONDARY OUTCOMES:
SUE (Subjective Units of Experience) Scale | 4 months
  The SUE (Subjective Experience Unit) scale evaluates the energy flow in the energy body. Emotions provide information about the state of the energy body. It is a simplified form of the stress table and measures the level of emotion experienced by the person. It was created by Hartman (2009) with the "Event Psychology" approach.
  The scores obtained on the SUE scale provide concrete and basic data about the current state of the person and after EFT, and show how there will be a change in this process. On the scale from "-10" to "+10", the person rates the anxiety or distress he feels. On this scale from -10 to +10; If the mood of the person is "-10", it is evaluated as very bad/negative, "0" as neutral, and "+10" as positive. Frustration, greatest pain, anxiety, fear or discomfort in the minds of -10 people is defined as the highest level of happiness, joy or feeling very well of the individual

CONTACTS AND LOCATIONS:
Overall Officials: Şule Ecevit Alpar, Phd, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No